CLINICAL TRIAL: NCT01429259
Title: An Open Label Study to Assess the Population Pharmacokinetics, Safety, and Practicality of Administering Meropenem as a Prolonged Infusion to Cystic Fibrosis Children Admitted With an Acute Pulmonary Exacerbation
Brief Title: Population Pharmacokinetics of Prolonged Infusion Meropenem in Cystic Fibrosis (CF) Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joseph Kuti (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor-Investigator, Joseph Kuti, Associate Director, Center for Anti-Infective Research and Development, Hartford Hospital
Organization: Hartford Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUTI003498HE
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-02

CONDITIONS: Cystic Fibrosis; Pneumonia; Pseudomonas Aeruginosa Infection
Keywords: Cystic Fibrosis; Acute Pulmonary Exacerbations; Pseudomonas aeruginosa
MeSH Terms: conditions — Cystic Fibrosis; Pneumonia; Pseudomonas Infections | interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Meropenem 3 hour prolonged infusion (Experimental): All 30 participants will receive meropenem as a 3 hour infusion.
  Interventions: Drug: meropenem

INTERVENTIONS:
Drug: meropenem — meropenem 40mg/kg total body weight will be administered every 8 hours. Each infusion will be infused as a 3 hour infusion.
  Other Names: Merrem

SUMMARY:
This study will determine the concentrations of the antibiotic meropenem when administered as a 3 hour prolonged infusion in children with cystic fibrosis who are hospitalized with an acute pulmonary exacerbation. Safety and practicality of administering meropenem as a 3 hour infusion will be measured.

DETAILED DESCRIPTION:
This study will be conducted at 7 pediatric hospitals in the United States (Columbia University Medical Center, New York, New York; University of North Carolina, Chapel Hill, North Carolina; St. Christopher's Hospital for Children, Philadelphia, Pennsylvania, Connecticut Children's Medical Center, Hartford, Connecticut, Riley Hospital for Children, Indianapolis, Indiana, Nationwide Hospital for Children, Columbus, Ohio, and Children's Medical Center, Dallas, Texas). Cystic Fibrosis children (age 6-17 years) admitted to one of these enrolling sites with an acute exacerbation of his or her pulmonary infection who require antibiotic therapy with meropenem will be eligible. Meropenem will be administered as a 3 hour prolonged infusion and blood concentrations will be measured to determine the population pharmacokinetics in 30 patients, the safety of prolonged infusion meropenem, and the practicality as measured be treatment burden using a questionaire. The population pharmacokinetic model developed will be utilized to determine the optimal dose of meropenem to administer to children with Cystic Fibrosis, and define an exposure response relationship for the drug in this population.

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis
* Hospitalized with acute pulmonary exacerbation
* Caused by Pseudomonas aeruginosa or other bacteria against which meropenem would be an appropriate antibiotic treatment

Exclusion Criteria:

* Known allergy to meropenem
* Require less than 3 days of meropenem in the hospital
* Require another systemic Beta-lactam antibiotic to treat a concomitant pathogen
* Known fungal or viral infection
* Females in their 2nd or 3rd trimester of pregnancy
* Moderate to severe renal dysfunction, as defined by a creatinine clearance less than 50 ml/min/1.73m2 (by use of Schwartz method)
* History of solid organ transplantation within previous 6 months
* Active or recent (within 30 days) participation in another antibiotic clinical trial

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Kuti, Pharm.D., Principal Investigator — Hartford Hospital
Locations (7):
- United States (7):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Riley Hospital for Children, Indianapolis, Indiana
  - Columbia University Medical Center Children's Hospital, New York, New York
  - University of North Carolina, North Carolina Children's Hospital, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Pettit RS, Neu N, Cies JJ, Lapin C, Muhlebach MS, Novak KJ, Nguyen ST, Saiman L, Nicolau DP, Kuti JL. Population pharmacokinetics of meropenem administered as a prolonged infusion in children with cystic fibrosis. J Antimicrob Chemother. 2016 Jan;71(1):189-95. doi: 10.1093/jac/dkv289. Epub 2015 Sep 27. PMID 26416780

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Meropenem 3 Hour Prolonged Infusion
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Enrolled participants receiving at least 3 doses of meropenem as a 3 hour prolonged infusion.
Arm/Group | Meropenem 3 Hour Prolonged Infusion
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.7 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Baseline Forced Expiratory Volume in 1st Second (FEV1) (% predicted) [Mean (Standard Deviation); unit: % predicted] | 58 (24)
Historical Best FEV1 (% predicted) [Mean (Standard Deviation); unit: % predicted] — The Historical Best FEV1 baseline measure estimates the baseline decline in pulmonary function of the population when not having an acute exacerbation. This value should be greater than the Baseline FEV1 thereby supporting that patients were having an acute pulmonary exacerbation at the start of the study.
  % predicted | 71 (25)

OUTCOME MEASURES:

1. Primary Outcome: Population Pharmacokinetics - Total Body Clearance
Description: Based on meropenem concentrations, the pharmacokinetics of the study population will be analyzed to determine each patient's total body clearance.
Time Frame: 8 hour dosing interval after 3rd meropenem dose
Measure: Mean (Standard Deviation); unit: L/hr/kg
Arm/Group | Meropenem 3 Hour Prolonged Infusion
Number analyzed (Participants) | 30
L/hr/kg | 0.36 (0.14)

2. Primary Outcome: Population Pharmacokinetics - Volume of Central Compartment
Description: Based on meropenem concentrations, the pharmacokinetics of the study population will be analyzed to determine each patient's volume of the central compartment.
Time Frame: During 8 hour dosing interval after 3rd meropenem dose
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Meropenem 3 Hour Prolonged Infusion
Number analyzed (Participants) | 30
L/kg | 0.21 (0.15)

3. Secondary Outcome: Safety
Description: This will be an intention to treat analysis of all 30 participants receiving meropenem as a 3 hour prolonged infusion. Participants will be monitored for any sign of symptom of adverse events throughout the course of the study. An adverse event will be defined as any pathologic or unintended change in the structure (signs), function (symptoms), or chemistry (laboratory values) of the body associated with the use of the study drug.
Time Frame: 14-21 days
Reporting Status: Not Posted

4. Secondary Outcome: Practicality of 3 Hour Prolonged Infusion
Description: This will be an intention to treat analysis of all 30 participants receiving meropenem as a 3 hour prolonged infusion. The Cystic Fibrosis Questionnaire-Revised (CFQ-R) will be utilized to assess patient or parent assessments of the burden of the prolonged infusion treatment. The CFQ-R will be administered at the beginning of the study and then within 7 days after completion of meropenem therapy.
Time Frame: 14-21 days
Reporting Status: Not Posted

5. Secondary Outcome: Meropenem Pharmacodynamics
Description: Meropenem exposures defined from the population model for each participant will be analyzed as a function of the isolated pathogens meropenem minimum inhibitory concentration (MIC) to define the exposure of meropenem associated with an absolute and relative percent change in the Forced Expiratory Volume (FEV1).
Time Frame: 14-21 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events collected from time of consent until completion of the study, which was 7-14 days after completion of meropenem prolonged infusion.
Description: Laboratory (chemistry, complete blood count, liver function tests, urinalysis) systematically collected at baseline and end of therapy. Other adverse events documented when reported by the participant or on findings during physical examination.
Arm/Group | Meropenem 3 Hour Prolonged Infusion
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 7/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meropenem 3 Hour Prolonged Infusion (N=30)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) — White Blood Cell count decreased from normal to 2.8 thousand cells/microliter; Absolute Neutrophil Count=1960; Hematocrit reduced to 30.2%; Platelets decreased to 39 thousand cells/microliter. This adverse event led to prolongation of hospital stay.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Meropenem 3 Hour Prolonged Infusion (N=30)
Leukocytosis (Blood and lymphatic system disorders) | 1
Thrombocythemia (Blood and lymphatic system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Fever (General disorders) | 2
C-Reactive Protein Elevation (Immune system disorders) | 3
Clostridium difficile Infection (Infections and infestations) | 2
Liver Function Test Abnormality (Hepatobiliary disorders) | 2 — Elevation in aspartate aminotransferase and alanine aminotransferase
Hyperbilirubinemia (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No